CLINICAL TRIAL: NCT03624608
Title: Evaluation of the Auryzon Family of Cartilage Processing Devices in the Optimization of Cartilaginous Reconstructions
Brief Title: Evaluation of the Auryzon Devices in the Optimization of Ear and Nose Reconstruction Procedures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment target not reached.
Sponsor: Reconstrata, LLC (Industry)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZN-001
Record Dates: First submitted 2018-07-22; First posted 2018-08-10 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Ear Deformities, Acquired; Ear; Deformity, Congenital; Microtia; Nose Deformity; Nose Deformities, Acquired; Nose; Deformity, Congenital; Nose; Deformity, Congenital, Bent or Squashed; Nose; Deformity, Syphilitic, Congenital; Nose; Deformity, Bone (Nose Cartilage); Nose; Deformity, Septum, Congenital; Nose; Deformity, Sinus (Wall), Congenital; Nose; Deformity, Syphilitic, Late (Etiology); Ear; Deformity, External; Ear; Deformity, Auricle, Ear, Acquired; Ear; Deformity, Auricle, Ear (Congenital)
MeSH Terms: conditions — Ear Deformities, Acquired; Congenital Abnormalities; Congenital Microtia; Nose Deformities, Acquired; Airway Obstruction; Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Auryzon-Processed Ear/Nose (Experimental): Patients in this category underwent reconstruction and implantation of a completed ear/nose cartilaginous graft that was processed using the AuryzoN device.
  Interventions: Device: AuryzoN Family of Devices

INTERVENTIONS:
Device: AuryzoN Family of Devices — The AuryzoN family of devices includes a longitudinal cartilage trimmer (DimensioN) and 2D shape carving machine with custom blades (AuryzoN).

SUMMARY:
This study evaluates the efficacy of the AuryzoN devices in the ear and nose reconstruction surgeries, both in terms of operative time and overall quality of reconstruction. Research participants will undergo reconstruction either using the AuryzoN device or through current methods (traditional manual processing) at the discretion of their surgeon prior to the start of surgery.

DETAILED DESCRIPTION:
The AuryzoN devices are a family of two (2) devices that, in conjunction, serve to process substrates of autologous-derived or cadaveric cartilage used in the reconstruction of various structures of the body, namely ear and nose. The devices are to be used in the operating room to cut and carve substrates of tissue into components, which are then assembled into the final ear or nose, that will then be implanted by the plastic surgeon into the appropriate area. This device family serves to replace the current step in this reconstructive procedure, which involves the time-consuming and error-prone process of manual cartilage processing.

Participants will be given the option to participate in the study. If the participants so choose, they will undergo ear or nose reconstruction using the AuryzoN devices or traditional manual processing at the discretion of their surgeon prior to the start of surgery. The following outcome measures will be measured: operative time, error rates, objective quality outcomes of reconstruction, subjective quality outcomes of reconstruction, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1-100 of sufficient health required to undergo ear/nose reconstruction under general anesthesia
* Pre-existing physical deformity of the ear, nose, or eyelid necessitating surgical reconstruction
* Sufficient autologous or cadaveric rib cartilage for use by the AuryzoN system for cartilage processing

Exclusion Criteria:

* Patients with ear/nose/eyelid deformities not requiring surgical correction
* Patients without sufficient rib cartilage for use by the AuryzoN system and those who do not desire cadaveric cartilage use
* Patients in poor health to undergo surgery under general anesthesia
* Patients whose desired ear/nose/eyelid exceeds the dimensions/shapes of those pre-fabricated blades used in the AuryzoN system

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Total cartilage processing time | Three years (until 2023)
  Total operative time spent by the surgeon preparing cartilage substrate into finished structures
Objective Quality of Reconstruction | Up to 1 year post-op (until 2023)
  An objective scoring system will be developed to score ears and noses based on anatomic accuracy, and reconstructed ears/noses will be scored using this system.
  Scoring system scale: The following metrics will be assessed by independent observers on a scale from 0-5, with 5 indicating perfect anatomic fidelity as compared to the patient's contralateral ear (or a model ear if no contralateral ear is available) or model nose and 0 indicating complete anatomical difference or loss of that structure.
  The following ear and nose subcomponents will be graded:
  Ear: Helix, antihelix, tragus, crus, anatomical proportion of all substrates as compared to each other substrate.
  Nose: Septum, alar cartilages, lateral cartilages, horizontal strut, anatomical proportion of all substrates as compared to each other substrate.

SECONDARY OUTCOMES:
Total operative time | Three years (until 2023)
  Total operative time by the surgeon performing the reconstructive surgery
Cartilage processing error rate | Three years (until 2023)
  Number of errors (defined as anatomic deviations) incurred during cartilaginous processing
Patient satisfaction | Up to 1 year post-op (until 2023)
  Subjective survey completed by patients asking about satisfaction with reconstruction
Subjective Quality of Reconstruction | Up to 1 year post-op (until 2023)
  Images of completed ear/nose reconstructions with the AuryzoN system will be presented to surgeons and lay-people to determine overall subjective quality of reconstruction

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Leto Barone, Principal Investigator — Reconstrata, LLC
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Leto Barone AA, Arun A, Samaha GJ, Shallal CC, Redett RJ, Steinberg JP. Design of a Novel Reproducible Cartilage-Sparing Autologous Technique for Microtia Repair. Facial Plast Surg Aesthet Med. 2021 May-Jun;23(3):224-229. doi: 10.1089/fpsam.2020.0457. Epub 2020 Nov 12. PMID 33185490